CLINICAL TRIAL: NCT00716144
Title: A Randomized, Evaluator-Blind, Placebo-Controlled, Parallel-Group Dose-Ranging Study of the Safety and Efficacy of Oral R115866 and R115866 Placebo in the Treatment of Plaque Psoriasis
Brief Title: Dose Ranging Study of the Safety and Efficacy of R115966 in Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BT0720-201-INT
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Results first posted 2018-01-29 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2017-05

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — R 115866

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Active Comparator): Talarozole 0.5 mg
  Interventions: Drug: Talarozole
- B (Active Comparator): Talarozole 1.0 mg
  Interventions: Drug: Talarozole
- C (Active Comparator): Talarozole 2.0 mg
  Interventions: Drug: Talarozole
- D (Placebo Comparator): Talarozole matching Placebo
  Interventions: Drug: Talarozole

INTERVENTIONS:
Drug: Talarozole — Oral Capsule Once Daily
  Other Names: Rambazole; R115866

SUMMARY:
Eligible subjects will be randomly assigned to one of three dose regimens of oral R115866 or placebo for the treatment of severe plaque psoriasis for 12 twelve weeks. The safety and efficacy of R115866 will be evaluated during the treatment period and the 8-week post treatment follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Plaque Psoriasis with PASI greater than or equal to 10
* Male or a female who was NOT of childbearing potential (i.e., post- menopausal for greater than 12 months or had a complete hysterectomy);

Exclusion Criteria:

* Spontaneously improving or rapidly deteriorating plaque psoriasis
* Guttate, pustular, erythrodermic, or other non-plaque form of psoriasis
* Subject was under treatment for a heart disorder or had a history of cardiovascular disease (excluding effectively controlled hypertension)
* Any acute psychiatric condition, including an increased risk for suicide attempt, based on medical and psychiatric history
* Previous use of a psoriasis vaccine or had participated in an investigational study of a psoriasis vaccine
* Previous use of systemic immunomodulatory therapy known to affect psoriasis and to typically decrease immune cell populations
* Previous use of any systemic immunomodulatory therapy known to affect psoriasis and NOT typically to decrease immune cell populations
* Previous use of any photo-therapy (including laser), photo-chemotherapy, or systemic psoriasis therapy (such as systemic corticosteroids, methotrexate, retinoids, or cyclosporine) within the previous four weeks
* Pregnant or a nursing mother
* Significant coexisting hepatic, renal, or bone marrow disease, hyperlipidemia, chronic pancreatitis, osteoporosis, cancer (except non-melanoma skin cancer), a positive test for human immunodeficiency virus (HIV), a history indicating adrenal cortex dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2006-06-01; Primary Completion 2007-05-01 (Actual); Study Completion 2007-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (22):
- Germany (6):
  - GSK Investigational Site, Augsburg
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Dresden
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Salzwedel
- GSK Investigational Site, Cork, Ireland
- Netherlands (2):
  - GSK Investigational Site, Maastricht
  - GSK Investigational Site, Nijmegen
- Russia (7):
  - GSK Investigational Site, Korolyov
  - GSK Investigational Site, Lipetsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Veliky Novgorod
  - GSK Investigational Site, Yaroslavl
- United Kingdom (6):
  - GSK Investigational Site, Aberdeen
  - GSK Investigational Site, Amersham
  - GSK Investigational Site, Coventry
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Norwich

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 176 participants were randomized into the study. This study was conducted at 25 centers located in Ireland, the United Kingdom, the Netherlands, Germany, and Russia from 19 June 2006 to 18 May 2007.
Pre-assignment Details: All participants were screened (Visit 1) two weeks prior to randomization (Visit 2) in order to evaluate their eligibility for entry into the trial. At Visit 1, participants signed an informed consent, provided their medical histories, reported their concomitant medication usages, and were evaluated against the inclusion/exclusion criteria.
Groups:
- Placebo: Eligible participants received R115866 matching placebo capsule orally, one capsule daily each morning with a meal for the 12 week treatment period.
- R115866 0.5 mg: Eligible participants received R115866 softgel capsule 0.5 milligram (mg) orally, one capsule daily each morning with a meal for the 12 week treatment period.
- R115866 1.0 mg: Eligible participants received R115866 softgel capsule 1.0 mg orally, one capsule daily each morning with a meal for the 12 week treatment period.
- R115866 2.0 mg: Eligible participants received R115866 softgel capsule 2.0 mg orally, one capsule daily each morning with a meal for the 12 week treatment period.
Period: Overall Study
Arm/Group | Placebo | R115866 0.5 mg | R115866 1.0 mg | R115866 2.0 mg
Started | 41 | 45 | 45 | 45
Completed | 32 | 38 | 33 | 33
Not Completed | 9 | 7 | 12 | 12
Not completed — Withdrawal by Subject | 4 | 2 | 6 | 6
Not completed — Lost to Follow-up | 2 | 2 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Non-compliance | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 2 | 2
Not completed — Intercurrent illness | 0 | 0 | 1 | 0
Not completed — Withdrew consent, allowed use of data | 0 | 0 | 1 | 0
Not completed — Adverse event: left foot pain | 0 | 1 | 0 | 0
Not completed — Clinical Depression | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- R115866 0.5 mg: Eligible participants received R115866 softgel capsule 0.5 mg orally, one capsule daily each morning with a meal for the 12 week treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo | R115866 0.5 mg | R115866 1.0 mg | R115866 2.0 mg | Total
Number analyzed (Participants) | 41 | 45 | 45 | 45 | 176
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.9 (12.3) | 42.3 (13.3) | 47.3 (11.5) | 48.2 (12.4) | NA (NA) — Age totals (mean and SD) were not provided in CSR. The raw data for this study is no longer available in any of our statistical systems, despite a thorough search. We are unable to supply this total data as typically required.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 3 | 6 | 15
  Male | 37 | 43 | 42 | 39 | 161
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 40 | 45 | 44 | 45 | 174
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Psoriasis Area Severity Index (PASI)75 Success at Visit 6
Description: PASI75 success at Visit 6 was defined as number of participants who achieved at least 75% reduction in PASI scores at Visit 6 compared to Visit 2 (Baseline). The PASI score was determined through evaluation of body surface area (BSA) covered by plaque psoriasis in four regions (head/neck, upper extremities, trunk and lower extremities). This assessment included a combination of both degree of involvement (assessed as per the % of affected body area using a 7-point scale that ranged as 0 (0% involvement), 1 = 1-9%, 2 = 10-29%, 3 = 30-49%, 4 = 50-69%, 5 = 70-89% and 6 = 90-100%) and severity (evaluated individually using a 5-point scale that ranged as 0 = No evidence of sign, 1 = slight evidence of sign, 2 = moderate evidence of sign, 3 = marked evidence of sign and 4 = very marked, most severe evidence of sign) of erythema, induration and desquamation in each of the same four regions. PASI score ranged from 0 to 72 in 0.1-unit intervals; higher scores indicating worse psoriasis.
Time Frame: Week 12 (Visit 6)
Population: Modified Intent-to-Treat (MITT) population. MITT population comprised of all randomized participants who took study medication and provided post-Visit 2 efficacy data (i.e., had one on-therapy follow-up visit).
Measure: Number; unit: Participants
Arm/Group | Placebo | R115866 0.5 mg | R115866 1.0 mg | R115866 2.0 mg
Number analyzed (Participants) | 41 | 45 | 45 | 45
Participants | 4 | 7 | 4 | 5
Statistical Analysis 1: Comparison: Placebo vs R115866 0.5 mg vs R115866 1.0 mg vs R115866 2.0 mg; Test type: Superiority or Other; p = 0.884, Cochran-Armitage Trend Test

2. Secondary Outcome: PASI50 Success (the Reduction in PASI Score at Each Visit of at Least 50 Percent Relative to Visit 2) at Each Post Baseline Visit
Description: PASI50 success was defined as number of participants who achieved at least 50% reduction in PASI scores at each post baseline visit (Visit 3 to 8) compared to Visit 2 (Baseline). The PASI score was determined through evaluation of BSA covered by plaque psoriasis in four regions (head/neck, upper extremities, trunk and lower extremities). This assessment included a combination of both degree of involvement (assessed as per the % of affected body area using a 7-point scale that ranged as 0 (0% involvement), 1 = 1-9%, 2 = 10-29%, 3 = 30-49%, 4 = 50-69%, 5 = 70-89% and 6 = 90-100%) and severity (evaluated individually using a 5-point scale that ranged as 0 = No evidence of sign, 1 = slight evidence of sign, 2 = moderate evidence of sign, 3 = marked evidence of sign and 4 = very marked, most severe evidence of sign) of erythema, induration and desquamation in each of the same four regions. PASI score ranged from 0 to 72 in 0.1-unit intervals; higher scores indicating worse psoriasis.
Time Frame: Week 1 to Week 20 (Visit 3 to Visit 8)
Population: MITT population.
Measure: Number; unit: Participants
Arm/Group | Placebo | R115866 0.5 mg | R115866 1.0 mg | R115866 2.0 mg
Number analyzed (Participants) | 41 | 45 | 45 | 45
Participants
  Visit 3 | 0 | 0 | 0 | 0
  Visit 4 | 2 | 0 | 1 | 1
  Visit 5 | 7 | 9 | 8 | 11
  Visit 6 | 8 | 18 | 18 | 19
  Visit 7 | 11 | 18 | 17 | 21
  Visit 8 | 15 | 16 | 18 | 24
Statistical Analysis 1: Comparison: Placebo vs R115866 0.5 mg vs R115866 1.0 mg vs R115866 2.0 mg; At Visit 3; Test type: Superiority or Other; p = 1.000, Cochran-Armitage Trend Test
Statistical Analysis 2: Comparison: Placebo vs R115866 0.5 mg vs R115866 1.0 mg vs R115866 2.0 mg; At Visit 4; Test type: Superiority or Other; p = 0.604, Cochran-Armitage Trend Test
Statistical Analysis 3: Comparison: Placebo vs R115866 0.5 mg vs R115866 1.0 mg vs R115866 2.0 mg; At Visit 5; Test type: Superiority or Other; p = 0.463, Cochran-Armitage Trend Test
Statistical Analysis 4: Comparison: Placebo vs R115866 0.5 mg vs R115866 1.0 mg vs R115866 2.0 mg; At Visit 6; Test type: Superiority or Other; p = 0.042, Cochran-Armitage Trend Test
Statistical Analysis 5: Comparison: Placebo vs R115866 0.5 mg vs R115866 1.0 mg vs R115866 2.0 mg; At Visit 7; Test type: Superiority or Other; p = 0.034, Cochran-Armitage Trend Test
Statistical Analysis 6: Comparison: Placebo vs R115866 0.5 mg vs R115866 1.0 mg vs R115866 2.0 mg; At Visit 8; Test type: Superiority or Other; p = 0.019, Cochran-Armitage Trend Test

3. Secondary Outcome: Investigator's Global Assessment (IGA) at Each Post Baseline Visit
Description: The IGA was used to assess the overall severity of a participant's plaque psoriasis at a particular time point and the evaluation took into consideration the three individual characteristics of plaque psoriasis (scaling, plaque elevation, and erythema). The IGA was recorded using a scale that ranged from 0 (clear), 1 = almost clear, 2 = mild, 3 = moderate to 4 (severe) in whole-unit increments; higher scores indicating worse psoriasis. Investigators did not refer to previous evaluations when conducting the IGA assessment. At every study visit, the investigator evaluated each participant's plaque psoriasis and recorded the one integer grade that best described the average, overall severity of the condition. Investigators were trained not to refer to previous assessments of the IGA, and not to base the IGA scores on any component of the PASI. Individual body regions were not assessed (as in the PASI), but rather a global evaluation for each participant at each visit was determined.
Time Frame: Week 1 to Week 20 (Visit 3 to Visit 8)
Population: MITT population. Only those participants available at the specified time points were analyzed. Different participants may have been analyzed at different time points; thus, the overall number of participants analyzed reflects everyone in the MITT Population.
Measure: Number; unit: Participants
Arm/Group | Placebo | R115866 0.5 mg | R115866 1.0 mg | R115866 2.0 mg
Number analyzed (Participants) | 41 | 45 | 45 | 45
Participants
  Clear; Visit 3 | 0 | 0 | 0 | 0
  Almost clear; Visit 3 | 0 | 0 | 0 | 0
  Mild; Visit 3 | 8 | 7 | 12 | 15
  Moderate; Visit 3 | 27 | 31 | 30 | 25
  Severe; Visit 3 | 6 | 7 | 3 | 5
  Clear; Visit 4 | 0 | 0 | 0 | 0
  Almost clear; Visit 4 | 0 | 0 | 0 | 0
  Mild; Visit 4 | 15 | 14 | 19 | 18
  Moderate; Visit 4 | 22 | 28 | 22 | 24
  Severe; Visit 4 | 4 | 3 | 4 | 3
  Clear; Visit 5 | 0 | 0 | 0 | 0
  Almost clear; Visit 5 | 3 | 2 | 3 | 6
  Mild; Visit 5 | 15 | 21 | 15 | 18
  Moderate; Visit 5 | 21 | 21 | 25 | 18
  Severe; Visit 5 | 2 | 1 | 2 | 3
  Clear; Visit 6 | 1 | 0 | 0 | 0
  Almost clear; Visit 6 | 3 | 9 | 6 | 11
  Mild; Visit 6 | 18 | 24 | 20 | 22
  Moderate; Visit 6 | 17 | 12 | 18 | 9
  Severe; Visit 6 | 2 | 0 | 1 | 3
  Clear; Visit 7: number analyzed (Participants) | 34 | 39 | 35 | 36
  Clear; Visit 7 | 0 | 0 | 0 | 0
  Almost clear; Visit 7: number analyzed (Participants) | 34 | 39 | 35 | 36
  Almost clear; Visit 7 | 5 | 11 | 8 | 14
  Mild; Visit 7: number analyzed (Participants) | 34 | 39 | 35 | 36
  Mild; Visit 7 | 15 | 19 | 16 | 14
  Moderate; Visit 7: number analyzed (Participants) | 34 | 39 | 35 | 36
  Moderate; Visit 7 | 13 | 8 | 11 | 8
  Severe; Visit 7: number analyzed (Participants) | 34 | 39 | 35 | 36
  Severe; Visit 7 | 1 | 1 | 0 | 0
  Clear; Visit 8: number analyzed (Participants) | 35 | 38 | 34 | 35
  Clear; Visit 8 | 1 | 0 | 2 | 2
  Almost clear; Visit 8: number analyzed (Participants) | 35 | 38 | 34 | 35
  Almost clear; Visit 8 | 6 | 6 | 9 | 15
  Mild; Visit 8: number analyzed (Participants) | 35 | 38 | 34 | 35
  Mild; Visit 8 | 15 | 21 | 10 | 10
  Moderate; Visit 8: number analyzed (Participants) | 35 | 38 | 34 | 35
  Moderate; Visit 8 | 10 | 10 | 12 | 8
  Severe; Visit 8: number analyzed (Participants) | 35 | 38 | 34 | 35
  Severe; Visit 8 | 3 | 1 | 1 | 0

4. Secondary Outcome: PASI75 at Each Post Baseline Visit Except Visit 6
Description: PASI75 success was defined as number of participants who achieved at least 75% reduction in PASI scores at each post baseline visit (Visit 3 to Visit 8) except Visit 6. The PASI score was determined through evaluation of BSA covered by plaque psoriasis in four regions (head/neck, upper extremities, trunk and lower extremities). This assessment included a combination of both degree of involvement (assessed as per the % of affected body area using a 7-point scale that ranged as 0 (0% involvement), 1 = 1-9%, 2 = 10-29%, 3 = 30-49%, 4 = 50-69%, 5 = 70-89% and 6 = 90-100%) and severity (evaluated individually using a 5-point scale that ranged as 0 = No evidence of sign, 1 = slight evidence of sign, 2 = moderate evidence of sign, 3 = marked evidence of sign and 4 = very marked, most severe evidence of sign) of erythema, induration and desquamation in each of the same four regions. PASI score ranged from 0 to 72 in 0.1-unit intervals; higher scores indicating worse psoriasis.
Time Frame: Week 1 to Week 20 (Visit 3 to Visit 8) except Week 12 (Visit 6)
Population: MITT population.
Measure: Number; unit: Participants
Arm/Group | Placebo | R115866 0.5 mg | R115866 1.0 mg | R115866 2.0 mg
Number analyzed (Participants) | 41 | 45 | 45 | 45
Participants
  Visit 3 | 0 | 0 | 0 | 0
  Visit 4 | 0 | 0 | 1 | 0
  Visit 5 | 4 | 0 | 2 | 5
  Visit 7: number analyzed (Participants) | 34 | 39 | 35 | 36
  Visit 7 | 5 | 8 | 6 | 7
  Visit 8: number analyzed (Participants) | 35 | 38 | 34 | 35
  Visit 8 | 6 | 7 | 10 | 13
Statistical Analysis 1: Comparison: Placebo vs R115866 0.5 mg vs R115866 1.0 mg vs R115866 2.0 mg; At Visit 3; Test type: Superiority or Other; p = 1.000, Cochran-Armitage Trend Test
Statistical Analysis 2: Comparison: Placebo vs R115866 0.5 mg vs R115866 1.0 mg vs R115866 2.0 mg; At Visit 4; Test type: Superiority or Other; p = 0.673, Cochran-Armitage Trend Test
Statistical Analysis 3: Comparison: Placebo vs R115866 0.5 mg vs R115866 1.0 mg vs R115866 2.0 mg; At Visit 5; Test type: Superiority or Other; p = 0.550, Cochran-Armitage Trend Test
Statistical Analysis 4: Comparison: Placebo vs R115866 0.5 mg vs R115866 1.0 mg vs R115866 2.0 mg; At Visit 7; Test type: Superiority or Other; p = 0.721, Cochran-Armitage Trend Test
Statistical Analysis 5: Comparison: Placebo vs R115866 0.5 mg vs R115866 1.0 mg vs R115866 2.0 mg; At Visit 8; Test type: Superiority or Other; p = 0.030, Cochran-Armitage Trend Test

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (nSAEs) were collected from Week 1 (Visit 3 [the first, post-randomization study visit]) to Week 20 (Visit 8 or early discontinuation), that is for 20 weeks.
Description: SAEs and nSAEs are reported for the MITT population.
Arm/Group | Placebo | R115866 0.5 mg | R115866 1.0 mg | R115866 2.0 mg
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/45 | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 1/41 | 1/45 | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 20/41 | 34/45 | 38/45 | 37/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | R115866 0.5 mg (N=45) | R115866 1.0 mg (N=45) | R115866 2.0 mg (N=45)
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | R115866 0.5 mg (N=45) | R115866 1.0 mg (N=45) | R115866 2.0 mg (N=45)
Coagulopathy (Blood and lymphatic system disorders) | 2 | 3 | 1 | 2
Dry eye (Eye disorders) | 1 | 3 | 6 | 3
Cheilitis (Gastrointestinal disorders) | 0 | 10 | 13 | 7
Dry mouth (Gastrointestinal disorders) | 2 | 2 | 3 | 1
Lip dry (Gastrointestinal disorders) | 1 | 9 | 8 | 12
Nasopharyngitis (Infections and infestations) | 1 | 5 | 2 | 1
Blood cholesterol increased (Investigations) | 1 | 1 | 3 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 3 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 3 | 0 | 5
Prothrombin time prolonged (Investigations) | 3 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 4
Depressive symptom (Psychiatric disorders) | 2 | 3 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 4 | 8 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 4 | 2 | 4
Psoriasis (Skin and subcutaneous tissue disorders) | 3 | 1 | 3 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 4 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.